CLINICAL TRIAL: NCT03176069
Title: Evaluation and Comparison of Women Pelvic Floor With and Without Sexual Dysfunction (Vaginismus)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Profa. Dra. Vera Lúcia dos Santos Alves, Associate Professor, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 51995515.4.0000.5479
Record Dates: First submitted 2016-05-12; First posted 2017-06-05 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-06

CONDITIONS: Vaginismus; Sexual Dysfunctions; Muscular Hypertonicity; Muscle Tone Poor
Keywords: Vaginismus; Muscle Tone; Sexual dysfunctions
MeSH Terms: conditions — Vaginismus; Muscle Hypertonia; Muscle Hypotonia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - women diagnosed with vaginismus (Active Comparator): All patients will be submitted to anamnesis, physical examination, examination of the pelvic floor. The algometry will be performed with patient will be lying in a supine position (belly up), with the pelvis in a neutral position, back at 45º and feet supported in stirrups, for the verification the perineal pain threshold.
  The available treatment tools are educational, behavioral and rehabilitating. The physiotherapeutic treatment will consist of the following features:
  Kinesiotherapy Manual therapy Electrotherapy (electric electrostimulation, ultrasound) Behavioral therapy
  Interventions: Other: The physiotherapeutic treatment
- Group B - women without a diagnosis of vaginismus (Active Comparator): All patients will be submitted to anamnesis, physical examination, examination of the pelvic floor. The algometry will be performed with patient will be lying in a supine position (belly up), with the pelvis in a neutral position, back at 45º and feet supported in stirrups, for the verification the perineal pain threshold.
  Interventions: Other: Evaluation and Comparison of women pelvic floor with and without sexual dysfunction

INTERVENTIONS:
Other: Evaluation and Comparison of women pelvic floor with and without sexual dysfunction — Pelvic floor muscles will also be evaluated by electromyographic biofeedback.
  Arms: Group B - women without a diagnosis of vaginismus
Other: The physiotherapeutic treatment — The available treatment tools are educational, behavioral and rehabilitating. The physiotherapeutic treatment will consist of the following features:
  * Kinesiotherapy
  * Manual therapy
  * Electrotherapy (electric electrostimulation, ultrasound)
  * Behavioral therapy
  Arms: Group A - women diagnosed with vaginismus

SUMMARY:
Sexuality is considered one of the pillars of quality of life, an integral part of the personality of each individual. Being a basic human being need, it cannot be separated from other aspects of life. For several centuries and until recently, sexuality was considered the "lower instincts" expression related only to the sexual act. Sex is associated with "reproduction" of the sexual energy. On the other hand, the exercise of sexuality includes various factors such as the building of the sensitivity between individuals like touch, dance, fantasy, look, etc. For a long time feminine sexuality was predominantly focused on procreation and has only recently been considered as an integral part of sexual and reproductive rights of women. Vaginismus is a female sexual dysfunction that affects the quality of sexual and psychosocial lives of women, influencing the quality of the couple's relationship. The scientific literature emphasizes the importance of the examination, diagnosis and physical therapy for this dysfunction, but until now there is no quantification or evaluation of the pelvic floor muscles for this group of women, which justifies the realization of this project.

DETAILED DESCRIPTION:
Psychosocial, cultural and relational factors, frequently influenced by a rigid education, have been related to the etiology of sexual difficulties. Women with stable partners who maintain an no consummated pattern of sexual intercourse (vaginismus) reveal a history of sexual life affected by these factors.

Vaginismus is a female sexual dysfunction that affects the quality of sexual and psychosocial lives of women. It may influence both the quality of the couple's relationship and the overall emotional and motivational state of people in their daily activities.

There is a concordance in the scientific literature that physiotherapy is of high importance in the treatment of vaginismus. The scientific literature presents some studies confirming its importance and highlighting the satisfactory results obtained at posttreatment of these dysfunctions.

Considering the impact of vaginismus in the sexual life of couples, as well as the relevance of the development of wide-ranging intervention models in the treatment of this disorder, it is appropriate to conduct this study in order to identify and recognize parameters of muscle tonus of women with and without a diagnosis of vaginismus and also to study the effectiveness of physiotherapy resources applied in the treatment of vaginismus.

Objectives

1. Evaluate and compare the pelvic floor musculature of women with and without a diagnosis of vaginismus, by algometry and perineal electromyographic biofeedback;
2. Evaluate and compare the parameters of muscle tonus of the pelvic floor by perineal electromyographic biofeedback in women with and without a diagnosis of vaginismus;
3. Evaluate the pelvic floor musculature of women diagnosed with vaginismus, through algometry and electromyographic biofeedback, after the physiotherapeutic treatment;
4. Evaluate the quality of sexual life and sexual function of women with and without a diagnosis of vaginismus;
5. Evaluate the quality of sexual life and sexual function of women diagnosed with vaginismus, after physiotherapeutic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Sexual orientation - heterosexual
* Be in a stable relationship for at least six months
* Present vaginismus
* Did not initiated and/or performed previous vaginismus treatment
* Elementary school level
* Be available for weekly attendance at ambulatory

Exclusion Criteria:

* Severe psychiatric illness (psychosis) or physical incapacity (previous or current)
* Vaginismus, whose characteristics suggest the need for surgical treatment
* Cognitive downgrade
* Absence of a stable relationship
* Partner with sexual dysfunction that prevents penetration
* Presence of genital prolapse

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Quality sex life | 3 months
  Female Sexual Function Index
Female Sexual Function | 3 months
  Sex Index - Female Version (QS-F)
Verification of female anxiety | 3 months
  Hamilton Anxiety Rating Scale (Ham-A)
Verification of female depression | 3 months
  Beck Depression Inventory (BDI)
Check Muscle Activity | 3 months
  Electromyographic biofeedback
Evaluation of Pain | 3 months
  Functional pain scale
Evaluation of Pain | 3 months
  Algometry

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Casa of Sao Paulo Medical School, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herbenick D, Schick V, Sanders SA, Reece M, Fortenberry JD. Pain experienced during vaginal and anal intercourse with other-sex partners: findings from a nationally representative probability study in the United States. J Sex Med. 2015 Apr;12(4):1040-51. doi: 10.1111/jsm.12841. Epub 2015 Feb 4. PMID 25648245
- [Background] Edenfield AL, Levin PJ, Dieter AA, Amundsen CL, Siddiqui NY. Sexual activity and vaginal topography in women with symptomatic pelvic floor disorders. J Sex Med. 2015 Feb;12(2):416-23. doi: 10.1111/jsm.12716. Epub 2014 Oct 8. PMID 25293781
- [Background] Rosenbaum TY. Physiotherapy treatment of sexual pain disorders. J Sex Marital Ther. 2005 Jul-Sep;31(4):329-40. doi: 10.1080/00926230590950235. PMID 16020150
- [Background] Rosenbaum T. Addressing anxiety in vivo in physiotherapy treatment of women with severe vaginismus: a clinical approach. J Sex Marital Ther. 2011;37(2):89-93. doi: 10.1080/0092623X.2011.547340. PMID 21400333
- [Background] van Lankveld JJ, ter Kuile MM, de Groot HE, Melles R, Nefs J, Zandbergen M. Cognitive-behavioral therapy for women with lifelong vaginismus: a randomized waiting-list controlled trial of efficacy. J Consult Clin Psychol. 2006 Feb;74(1):168-78. doi: 10.1037/0022-006X.74.1.168. PMID 16551154
- [Background] Addar MH. The unconsummated marriage: causes and management. Clin Exp Obstet Gynecol. 2004;31(4):279-81. PMID 15672966
- [Background] Lahaie MA, Boyer SC, Amsel R, Khalife S, Binik YM. Vaginismus: a review of the literature on the classification/diagnosis, etiology and treatment. Womens Health (Lond). 2010 Sep;6(5):705-19. doi: 10.2217/whe.10.46. PMID 20887170
- [Background] Aydin S, Arioglu Aydin C, Batmaz G, Dansuk R. Effect of vaginal electrical stimulation on female sexual functions: a randomized study. J Sex Med. 2015 Feb;12(2):463-9. doi: 10.1111/jsm.12788. Epub 2014 Dec 3. PMID 25470078
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Biswas A, Ratnam SS. Vaginismus and outcome of treatment. Ann Acad Med Singap. 1995 Sep;24(5):755-8. PMID 8579326
- [Background] Bortolami A, Vanti C, Banchelli F, Guccione AA, Pillastrini P. Relationship between female pelvic floor dysfunction and sexual dysfunction: an observational study. J Sex Med. 2015 May;12(5):1233-41. doi: 10.1111/jsm.12882. Epub 2015 Apr 8. PMID 25855126
- [Background] De Lorenzi DR, Saciloto B. [Factors related to frequency of sexual activity of postmenopausal women]. Rev Assoc Med Bras (1992). 2006 Jul-Aug;52(4):256-60. doi: 10.1590/s0104-42302006000400027. Portuguese. PMID 16967145
- [Background] Engman M, Wijma K, Wijma B. Long-term coital behaviour in women treated with cognitive behaviour therapy for superficial coital pain and vaginismus. Cogn Behav Ther. 2010;39(3):193-202. doi: 10.1080/16506070903571014. PMID 20390584
- [Background] Kingsberg S, Althof SE. Evaluation and treatment of female sexual disorders. Int Urogynecol J Pelvic Floor Dysfunct. 2009 May;20 Suppl 1:S33-43. doi: 10.1007/s00192-009-0833-x. PMID 19440781
- [Background] Lewis RW, Fugl-Meyer KS, Corona G, Hayes RD, Laumann EO, Moreira ED Jr, Rellini AH, Segraves T. Definitions/epidemiology/risk factors for sexual dysfunction. J Sex Med. 2010 Apr;7(4 Pt 2):1598-607. doi: 10.1111/j.1743-6109.2010.01778.x. PMID 20388160
- [Background] Melnik T, Hawton K, McGuire H. Interventions for vaginismus. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD001760. doi: 10.1002/14651858.CD001760.pub2. PMID 23235583
- [Background] Pereira VM, Arias-Carrion O, Machado S, Nardi AE, Silva AC. Sex therapy for female sexual dysfunction. Int Arch Med. 2013 Sep 26;6(1):37. doi: 10.1186/1755-7682-6-37. PMID 24066697
- [Background] Reissing ED, Binik YM, Khalife S, Cohen D, Amsel R. Vaginal spasm, pain, and behavior: an empirical investigation of the diagnosis of vaginismus. Arch Sex Behav. 2004 Feb;33(1):5-17. doi: 10.1023/B:ASEB.0000007458.32852.c8. PMID 14739686
- [Background] Reissing ED. Consultation and treatment history and causal attributions in an online sample of women with lifelong and acquired vaginismus. J Sex Med. 2012 Jan;9(1):251-8. doi: 10.1111/j.1743-6109.2011.02534.x. Epub 2011 Oct 24. PMID 22024357
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Segraves R, Balon R, Clayton A. Proposal for changes in diagnostic criteria for sexual dysfunctions. J Sex Med. 2007 May;4(3):567-580. doi: 10.1111/j.1743-6109.2007.00455.x. Epub 2007 Apr 13. PMID 17433086
- [Background] Seo JT, Choe JH, Lee WS, Kim KH. Efficacy of functional electrical stimulation-biofeedback with sexual cognitive-behavioral therapy as treatment of vaginismus. Urology. 2005 Jul;66(1):77-81. doi: 10.1016/j.urology.2005.01.025. PMID 15992873
- [Background] Sirakov M. [Vaginismus and our experience in treating this sexual problem]. Akush Ginekol (Sofiia). 2013;52(1):61-6. Bulgarian. PMID 23805463